CLINICAL TRIAL: NCT06514872
Title: Prevalence and Determinants of Home Accidents Among Turkish Older Men and Women
Brief Title: Home Accidents Among Turkish Older Men and Women
Status: Completed | Type: Observational
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Mevlana GÜL, Asst. Prof, Ataturk University
Other Study IDs: AtaturkUni1
Record Dates: First submitted 2024-06-25; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Age Problem
Keywords: Older individuals; Home accident; Discrete choice model; Binary logistic regression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Turkish older: The data obtained from individuals aged 60 and above were used in this study.
  Interventions: Other: prevalance and determinants of home accidents

INTERVENTIONS:
Other: prevalance and determinants of home accidents — home accidents among Turkish older
  Other Names: Turkish older

SUMMARY:
Background: Home accidents are a significant public health issue in developed and developing countries. The present study aims to identify the factors associated with home accidents among older individuals in Türkiye.

Methods: Microdata obtained from the Türkiye Health Survey conducted by the Turkish Statistical Institute (TUIK) in 2019 and 2022 were utilized in the present study. Binary logistic regression analysis was used to determine factors influencing home accidents.

DETAILED DESCRIPTION:
Home accidents are a significant public health issue in developed and developing countries. Home refers to where older individuals spend most of their daily time, thus increasing their likelihood of experiencing any accidents at home. Home accidents are more common among older individuals and can lead to serious health consequences. Individuals aged 65 and above are particularly at high risk of home accidents due to physical, psychological, and social impairments. Musculoskeletal problems and sensory and motor function loss in this group increase the risk of accidents. Home accidents are assumed to be unintentional and can range from minor injuries to fatalities. These accidents can occur within the home and in surrounding areas such as garages, gardens, terraces, and stairs. While unintentional home and recreational injuries pose a risk for individuals aged 85 and older, outdoor injuries also pose a risk for younger, older individuals.

ELIGIBILITY:
Inclusion Criteria:

* Older individuals are at risk for home accidents due to their developmental characteristics

Exclusion Criteria:

- healthy volunteers

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The research utilised microdata from the Türkiye Health Survey, published by the Turkish Statistical Institute (TUIK) in 2019 and 2022
Sampling Method: Probability Sample
Enrollment: 8225 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Factors contributing to home accidents among older individuals to ensure home safety | 2019-2022
  The research utilised microdata from the Türkiye Health Survey, published by the Turkish Statistical Institute (TUIK) in 2019 and 2022. The study's dependent variable is the occurrence of home accidents, measured by the question, "Have you experienced a home accident resulting in injury in the last 12 months? (Yes, No)." The independent variables of this study are gender, education level, marital status, employment status, general health status, presence of arthrosis, urinary incontinence, wearing glasses, experiencing difficulty in carrying or holding items, experiencing difficulty in affording health care services, and survey year.

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Alkan, Prof. Dr., Study Chair — Ataturk University
Locations (1):
- Mevlana Gul, Yakutiye, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bonnal L, Gámez GB, Favard P, Oros C. Who gets injured at home? Evidence from older people in France. Bulletin of Economic Research. 2023;75(2):450-75
- [Background] Altiparmak S, Horasan GD. Accident prevalence and accident associated risk factors among elderly people living in nursing homes in. Turkish Journal of Geriatrics-Turk Geriatri Dergisi. 2012;15(3):292-8.
- [Background] Yapici G, Kurt A, Öner S, Sasmaz T, Bugdayci R. Determination of the Home Accident Frequency and Related Factors Among the People Older than 65 Years Old Living in Mersin City Center, Turkey. Sage Open. 2019;9(2).
- [Background] Stalenhoef PA, Diederiks JP, Knottnerus JA, Kester AD, Crebolder HF. A risk model for the prediction of recurrent falls in community-dwelling elderly: a prospective cohort study. J Clin Epidemiol. 2002 Nov;55(11):1088-94. doi: 10.1016/s0895-4356(02)00502-4. PMID 12507672
- [Background] Şeker A, Gökhan K. Bir sosyal politika alanı olarak yaşlılık ve sosyal hizmet uygulamaları. Nüfusbilim Dergisi. 2018;40:7-30.
- [Background] TÜİK. Dünya Nüfus Günü. Ankara: Türkiye İstatistik Kurumu; 2023.
- [Background] Umutlu S, Epik MT. Türkiye'de yaşlı nüfus ve sosyal politika uygulamaları. Sosyal ve Beşerî Bilimler Dergisi. 2019;11(1):29-43
- [Background] Sahin H, Erkal S. Evaluation of home accidents and fall behaviors of elderly. Turkish Journal of Geriatrics-Turk Geriatri Dergisi. 2016;19(3):195-201.
- [Background] Saberian P, Farhoud AR, Hasani-Sharamin P, Moghaddami M, Keshvari F. Epidemiological Features of Injured Patients Examined by Tehran Emergency Medical Service Technicians. Adv J Emerg Med. 2019 Jun 25;3(4):e40. doi: 10.22114/ajem.v0i0.198. eCollection 2019 Fall. PMID 31633095
- [Background] Mikos M, Trybulska A, Czerw A. Falls - the socio-economic and medical aspects important for developing prevention and treatment strategies. Ann Agric Environ Med. 2021 Sep 16;28(3):391-396. doi: 10.26444/aaem/122409. Epub 2020 May 28. PMID 34558259
- [Background] Florence CS, Bergen G, Atherly A, Burns E, Stevens J, Drake C. Medical Costs of Fatal and Nonfatal Falls in Older Adults. J Am Geriatr Soc. 2018 Apr;66(4):693-698. doi: 10.1111/jgs.15304. Epub 2018 Mar 7. PMID 29512120
- [Background] Bergen G, Stevens MR, Burns ER. Falls and Fall Injuries Among Adults Aged >/=65 Years - United States, 2014. MMWR Morb Mortal Wkly Rep. 2016 Sep 23;65(37):993-998. doi: 10.15585/mmwr.mm6537a2. PMID 27656914
- [Background] Morrison A, Fan T, Sen SS, Weisenfluh L. Epidemiology of falls and osteoporotic fractures: a systematic review. Clinicoecon Outcomes Res. 2013;5:9-18. doi: 10.2147/CEOR.S38721. Epub 2012 Dec 28. PMID 23300349
- [Background] Tinetti ME, Speechley M, Ginter SF. Risk factors for falls among elderly persons living in the community. N Engl J Med. 1988 Dec 29;319(26):1701-7. doi: 10.1056/NEJM198812293192604. PMID 3205267
- [Background] Hopewell S, Adedire O, Copsey BJ, Boniface GJ, Sherrington C, Clemson L, Close JC, Lamb SE. Multifactorial and multiple component interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2018 Jul 23;7(7):CD012221. doi: 10.1002/14651858.CD012221.pub2. PMID 30035305
- [Background] Esechie A, Bhardwaj A, Masel T, Raji M. Neurocognitive sequela of burn injury in the elderly. J Clin Neurosci. 2019 Jan;59:1-5. doi: 10.1016/j.jocn.2018.10.089. Epub 2018 Nov 3. PMID 30401568
- [Background] Karam BS, Patnaik R, Murphy P, deRoon-Cassini TA, Trevino C, Hemmila MR, Haines K, Puzio TJ, Charles A, Tignanelli C, Morris R. Improving mortality in older adult trauma patients: Are we doing better? J Trauma Acute Care Surg. 2022 Feb 1;92(2):413-421. doi: 10.1097/TA.0000000000003406. PMID 34554138
- [Background] Adams SD, Holcomb JB. Geriatric trauma. Curr Opin Crit Care. 2015 Dec;21(6):520-6. doi: 10.1097/MCC.0000000000000246. PMID 26539925
- [Background] Banks SE, Lewis MC. Trauma in the elderly: considerations for anesthetic management. Anesthesiol Clin. 2013 Mar;31(1):127-39. doi: 10.1016/j.anclin.2012.11.004. Epub 2012 Dec 13. PMID 23351539
- [Background] Keall MD, Guria J, Howden-Chapman P, Baker MG. Estimation of the social costs of home injury: a comparison with estimates for road injury. Accid Anal Prev. 2011 May;43(3):998-1002. doi: 10.1016/j.aap.2010.11.027. Epub 2010 Dec 31. PMID 21376893
- [Background] Braubach M, Power A. Housing Conditions and Risk: Reporting on a European Study of Housing Quality and Risk of Accidents for Older People. Journal of Housing for the Elderly. 2011;25(3):288-305.
- [Background] TurkStat. Türkiye Sağlık Araştırması (Turkey Health Survey) Ankara; 2022.
- [Background] Anderson LK, Lane K. Characteristics of falls and recurrent falls in residents of an aging in place community: A case-control study. Appl Nurs Res. 2020 Feb;51:151190. doi: 10.1016/j.apnr.2019.151190. Epub 2019 Oct 5. PMID 31734004
- [Background] Anderson PA, Magaziner JS, Mendelson DA, Switzer JA. Own the Fall: AOA Critical Issues. J Bone Joint Surg Am. 2021 Oct 20;103(20):e82. doi: 10.2106/JBJS.20.02254. PMID 34191752
- [Background] Moncatar TJR, Nakamura K, Siongco KL, Rahman M, Seino K. Prevalence and Determinants of Self-Reported Injuries among Community-Dwelling Older Adults in the Philippines: A 10-Year Pooled Analysis. Int J Environ Res Public Health. 2020 Jun 18;17(12):4372. doi: 10.3390/ijerph17124372. PMID 32570797
- [Background] Piffer S, Demonti S, Ramponi C, Giustini M, Pitidis A. Home accidents in the province of Trento. Ten years of observations regarding admissions to the emergency and first aid department. Ann Ig. 2021 Mar-Apr;33(2):152-162. doi: 10.7416/ai.2021.2421. PMID 33570087
- [Background] Romli MH, Tan MP, Mackenzie L, Lovarini M, Suttanon P, Clemson L. Falls amongst older people in Southeast Asia: a scoping review. Public Health. 2017 Apr;145:96-112. doi: 10.1016/j.puhe.2016.12.035. Epub 2017 Jan 21. PMID 28359399
- [Background] Sotoudeh GR, Mohammadi R, Mosallanezhad Z, Viitasara E, Soares JJF. A population study on factors associated with unintentional falls among Iranian older adults. BMC Geriatr. 2023 Dec 15;23(1):860. doi: 10.1186/s12877-023-04571-0. PMID 38102576
- [Background] van Schoor NM, Dennison E, Castell MV, Cooper C, Edwards MH, Maggi S, Pedersen NL, van der Pas S, Rijnhart JJM, Lips P, Deeg DJH; EPOSA research group. Clinical osteoarthritis of the hip and knee and fall risk: The role of low physical functioning and pain medication. Semin Arthritis Rheum. 2020 Jun;50(3):380-386. doi: 10.1016/j.semarthrit.2020.02.006. Epub 2020 Feb 19. PMID 32199610
- [Background] Alkan Ö, Güney E. Investigation of factors that affect the frequency of alcohol use of employees in Turkey. Journal of Substance Use. 2021;26(5):468-74.
- [Background] Mato ML, Acerbo FY, Lema R. Gender roles in the distribution of housework related to food. Revista De Salud Publica-Cordoba. 2022;27(1):88-103.
- [Background] Kerman KT, Betrus P. What makes a man a
- [Background] Jalali MT, Sarikhani Y, Askarian F, Marzaleh MA, Najibi SM, Delavari S. Factors facilitating and inhibiting the social participation of the elderly in health-oriented activities in Shiraz, Southern Iran. BMC Geriatr. 2023 Mar 27;23(1):175. doi: 10.1186/s12877-023-03892-4. PMID 36973677
- [Background] Demir Y. Eğitim, sağlık ve ar-ge harcamaları ile ekonomik büyüme arasındaki ilişkinin ARDL sınır testi ile belirlenmesi. MANAS Sosyal Araştırmalar Dergisi. 2021;10(3):1758-70.
- [Background] Ravindran RM, Kutty VR. Risk Factors for Fall-Related Injuries Leading to Hospitalization Among Community-Dwelling Older Persons: A Hospital-Based Case-Control Study in Thiruvananthapuram, Kerala, India. Asia Pac J Public Health. 2016 Jan;28(1 Suppl):70S-76S. doi: 10.1177/1010539515611229. Epub 2015 Oct 12. PMID 26463576
- [Background] Duan Y, Peiris DLIHK, Yang M, Liang W, Baker JS, Hu C, Shang B. Lifestyle Behaviors and Quality of Life Among Older Adults After the First Wave of the COVID-19 Pandemic in Hubei China. Front Public Health. 2021 Dec 10;9:744514. doi: 10.3389/fpubh.2021.744514. eCollection 2021. PMID 34957009
- [Background] Rapp K, Pfeiffer K. Depression, osteoporosis, falls and fractures. Osteologie. 2019;28(4):246-51.
- [Background] Lin XZ, Meng RL, Peng DD, Li C, Zheng XY, Xu HF, Xu XJ, Lin LF. Cross-sectional study on prevalence and risk factors for falls among the elderly in communities of Guangdong province, China. BMJ Open. 2022 Nov 14;12(11):e062257. doi: 10.1136/bmjopen-2022-062257. PMID 36375979
- [Background] Hirono T, Takeda R, Nishikawa T, Okudaira M, Kunugi S, Yoshiko A, Ueda S, Yoshimura A, Watanabe K. Motor unit firing patterns in older adults with low skeletal muscle mass. Arch Gerontol Geriatr. 2024 Jan;116:105151. doi: 10.1016/j.archger.2023.105151. Epub 2023 Aug 1. PMID 37544147
- [Background] Byun M, Kim J, Kim M. Physical and Psychological Factors Affecting Falls in Older Patients with Arthritis. Int J Environ Res Public Health. 2020 Feb 9;17(3):1098. doi: 10.3390/ijerph17031098. PMID 32050468
- [Background] Auais M, Alvarado B, Guerra R, Curcio C, Freeman EE, Ylli A, Guralnik J, Deshpande N. Fear of falling and its association with life-space mobility of older adults: a cross-sectional analysis using data from five international sites. Age Ageing. 2017 May 1;46(3):459-465. doi: 10.1093/ageing/afw239. PMID 28043980
- [Background] Liu M, Hou T, Li Y, Sun X, Szanton SL, Clemson L, Davidson PM. Fear of falling is as important as multiple previous falls in terms of limiting daily activities: a longitudinal study. BMC Geriatr. 2021 Jun 7;21(1):350. doi: 10.1186/s12877-021-02305-8. PMID 34098904
- [Background] Barros L, Carvalhais A, Brochado G, Ferreira M. Functional ability and urinary incontinence in elderly women. European Journal of Public Health. 2019;29(Supplement_1):ckz034. 27.
- [Background] Mehta J, Czanner G, Harding S, Newsham D, Robinson J. Visual risk factors for falls in older adults: a case-control study. BMC Geriatr. 2022 Feb 17;22(1):134. doi: 10.1186/s12877-022-02784-3. PMID 35177024
- [Background] Moon BY, Choi JH, Yu DS, Kim SY. Effect of induced hyperopia on fall risk and Fourier transformation of postural sway. PeerJ. 2019 Dec 20;7:e8329. doi: 10.7717/peerj.8329. eCollection 2019. PMID 31879576
- [Background] Tieland M, Trouwborst I, Clark BC. Skeletal muscle performance and ageing. J Cachexia Sarcopenia Muscle. 2018 Feb;9(1):3-19. doi: 10.1002/jcsm.12238. Epub 2017 Nov 19. PMID 29151281
- [Background] Iamtrakul P, Chayphong S, Jomnonkwao S, Ratanavaraha V. The Association of Falls Risk in Older Adults and Their Living Environment: A Case Study of Rural Area, Thailand. Sustainability. 2021;13(24).
- [Result] Ferrante P, Marinaccio A, Iavicoli S. Home injuries in Italy: patterns of injury and the most exposed people. Int J Inj Contr Saf Promot. 2013;20(1):36-41. doi: 10.1080/17457300.2012.663761. Epub 2012 Mar 2. PMID 22385149
- [Result] Martin-Espinosa NM, Piriz-Campos RM, Cordeiro R, Munoz Bermejo L, Casado Verdjo I, Postigo Mota S. [SAFETY IN THE ELDERLY: HOME ACCIDENTS]. Rev Enferm. 2016 May;39(5):62-7. Spanish. PMID 27405149
- [Result] Samanci Tekin Ç, Kara F. Incidence of home accidents in 65 years of age and older individuals and related factors. Turkish Journal of Geriatrics-Turk Geriatri Dergisi. 2019;22(1):38-47.
- [Result] Spano G, O Caffo A, Bosco A. Cognitive functioning, subjective memory complaints and risky behaviour predict minor home injuries in elderly. Aging Clin Exp Res. 2018 Aug;30(8):985-991. doi: 10.1007/s40520-017-0858-9. Epub 2017 Nov 27. PMID 29181769

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT06514872/Prot_SAP_000.pdf